CLINICAL TRIAL: NCT02706405
Title: A Phase 1b Study of JCAR014, Autologous T Cells Engineered to Express a CD19-Specific Chimeric Antigen Receptor, in Combination With Durvalumab (MEDI4736) for Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: JCAR014 and Durvalumab in Treating Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry); MedImmune LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexandre Hirayama, Research Associate, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9457; NCI-2015-02286 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9457 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); R01CA136551 (NIH); RG6616001 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-02-24; First posted 2016-03-11 (Estimated); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma
Keywords: PD-L1; immunotherapy; non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; durvalumab; Immunoglobulin G; Disulfides; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group I (JCAR014, durvalumab) Early - Dose Level 2 (Experimental): Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - early: start durvalumab no earlier than 7 days after JCAR014.
  Group 1 Dose Level 2 is 750 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine
- Group I (JCAR014, durvalumab) Late- Dose Level 1 (Experimental): Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - late: start durvalumab no earlier than 21 days after JCAR014
  Group 1 Dose Level 1 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
  .
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine
- Group I (JCAR014, durvalumab) Late - Dose Level 2 (Experimental): Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - late: start durvalumab no earlier than 21 days after JCAR014
  Group 1 Dose Level 2 is 750 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine
- Group II (durvalumab, JCAR014) - Dose Level 1 (Experimental): Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 1 is 7.5 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine
- Group II (durvalumab, JCAR014) - Dose Level 2 (Experimental): Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 2 is 22.5 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine
- Group II (durvalumab, JCAR014) - Dose Level 3 (Experimental): Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 3 is 75 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine
- Group II (durvalumab, JCAR014) - Dose Level 4 (Experimental): Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 4 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine
- Group II (durvalumab, JCAR014) - Dose Level 5 (Experimental): Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 5 is 750 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Interventions: Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014; Drug: Cyclophosphamide; Biological: Durvalumab; Drug: Fludarabine

INTERVENTIONS:
Biological: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014 — Given IV
  Other Names: Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ CM T-lymphocytes JCAR014; JCAR014
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Fludarabine — Given IV
  Other Names: 2-Fluorovidarabine; Fluradosa

SUMMARY:
This phase Ib trial studies whether anti-CD19-chimeric antigen receptor (CAR) lentiviral vector-transduced autologous T cells (JCAR014) and durvalumab are safe in combination and can work together in treating patients with non-Hodgkin lymphoma that has returned after a period of improvement (relapsed) or has not responded to previous treatment (refractory). JCAR014 is made of each patient's immune cells (T cells) that have a new gene added to them in a laboratory, which programs them to kill lymphoma cells. Durvalumab is a type of drug called a monoclonal antibody, targeted to PD-L1 that may help immune cells attack cancer cells more effectively and thus help JCAR014 work better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of JCAR014 in combination with durvalumab in adult patients with relapsed/refractory (R/R) B-cell non-Hodgkin lymphoma (NHL).

II. To determine the maximum tolerated dose (MTD) of durvalumab in combination with JCAR014.

III. To characterize the pharmacokinetic (PK) profile of JCAR014.

SECONDARY OBJECTIVES:

I. To assess the antitumor activity of JCAR014 in combination with durvalumab in R/R B-cell NHL.

II. To estimate the duration of response (DOR), progression-free survival (PFS), and overall survival (OS) in patients treated with JCAR014 in combination with durvalumab.

III. To characterize the PK profile of durvalumab. IV. To assess the immunogenicity of JCAR014 and durvalumab.

EXPLORATORY OBJECTIVE:

I. To assess the pharmacodynamic effects of JCAR014 and durvalumab in blood and within the tumor.

OUTLINE: This is a dose-escalation study of durvalumab administered with a single fixed dose of JCAR014. Patients are assigned to 1 of 2 treatment arms, listed as Groups 1 and 2 below.

LYMPHODEPLETING CHEMOTHERAPY: All patients receive cyclophosphamide and fludarabine intravenously (IV) for 3 days starting approximately on day -5 or day -4.

GROUP I: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 30 days for 30 months, every 3 months for 12 months, then periodically for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR SCREENING:

* Relapsed or refractory diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS); high grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements; primary mediastinal B-cell lymphoma (PMBCL); or DLBCL transformed from indolent histology with one of the following:

  * Persistent disease after first-line chemo-immunotherapy
  * Relapse after first-line chemo-immunotherapy and not eligible for autologous hematopoietic stem cell transplant (HCT)
  * Relapse or persistent disease after at least two lines of therapy or after autologous HCT
* Ability to understand and provide informed consent

INCLUSION CRITERIA FOR LEUKAPHERESIS AND PRE-THERAPY EVALUATION:

* Screening evaluation appropriate for leukapheresis and T-cell collection
* Evidence of CD19 expression on any prior or current tumor specimen or a high likelihood of CD19 expression based on disease histology

INCLUSION CRITERIA FOR LYMPHODEPLETION CHEMOTHERAPY, JCAR014 AND DURVALUMAB:

* Successful collection of T cells for JCAR014 manufacturing
* Documentation of CD19 expression on any prior or current tumor biopsy
* Internal review of histology
* Detectable positron emission tomography (PET)-positive disease
* Karnofsky performance status >= 60%
* Assessed by the investigator to have adequate bone marrow function to receive lymphodepleting conditioning chemotherapy
* Serum creatinine < 1.5 x age-adjusted upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN and total bilirubin =< 2 x ULN
* Adequate pulmonary function, defined as Common Terminology Criteria for Adverse Events (CTCAE) grade =< 1 dyspnea and oxygen saturation (SaO2) >= 92% on room air; patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing and must have a forced expiratory volume in 1 second (FEV1) >= 50% of predicted value or diffusing capacity of the lung for carbon monoxide (DLCO; corrected) >= 40% of predicted value
* Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) >= 35% as assessed by echocardiogram (ECHO) or multiple uptake gated acquisition (MUGA)
* Women of reproductive potential (defined as all women physiologically capable of becoming pregnant) must agree to use suitable methods of contraception for 90 days after the last dose of study therapy (durvalumab or JCAR014)
* Males who have partners of reproductive potential must agree to use an effective barrier contraceptive method for 90 days after the last dose of study therapy (durvalumab or JCAR014)

Exclusion Criteria:

EXCLUSION CRITERIA FOR SCREENING:

* Subjects with known active central nervous system (CNS) involvement by malignancy; subjects with prior CNS disease that has been effectively treated will be eligible if treatment was completed at least 3 months prior to enrollment and there is no evidence of disease or stable abnormalities on repeat imaging
* Planned use of corticosteroids (> 10 mg/day prednisone or equivalent) or other systemic immunosuppression within 4 days prior to leukapheresis; topical and/or inhaled steroids are permitted
* Prior treatment with any CD19 CAR T-cell therapy
* Prior allogeneic HCT
* Known active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection
* Pregnant or breastfeeding women
* Known exclusion criteria for leukapheresis, JCAR014, or durvalumab therapy

EXCLUSION CRITERIA FOR LEUKAPHERESIS AND PRE-THERAPY EVALUATION:

* Subjects with known active central nervous system (CNS) involvement by malignancy; subjects with prior CNS disease that has been effectively treated will be eligible if treatment was completed at least 3 months prior to enrollment and there is no evidence of disease or stable abnormalities on repeat imaging
* Prior treatment with programmed cell death (PD)-1, PD-ligand (L)1, cytotoxic T lymphocyte-associated protein 4 (CTLA 4) targeted therapy, or tumor necrosis factor receptor superfamily (TNFRSF) agonists including CD134 (OX40), CD27, CD137 (4-1BB), and CD357 (glucocorticoid-induced tumor necrosis factor receptor family-related protein [GITR])
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., ulcerative colitis, Crohn's disease], celiac disease, or other serious chronic gastrointestinal conditions associated with diarrhea; autoimmune vasculitis; systemic lupus erythematosus; Wegener syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis, hypophysitis, uveitis, etc.) within 3 years prior to the planned start of treatment; the following are exceptions to this criterion:

  * Vitiligo
  * Alopecia
  * Hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Psoriasis not requiring systemic treatment
  * Other conditions considered to be low risk of serious deterioration by the principal investigator (PI)
* History of any one of the following cardiovascular conditions within the past 6 months: class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, or unstable angina; history of other clinically significant cardiac disease that, in the opinion of the PI or designee, is a contraindication to lymphodepleting chemotherapy, JCAR014 infusion, or durvalumab infusion is also excluded
* History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, or psychosis; history of other organic brain syndrome that in the opinion of the PI or designee is a contraindication to lymphodepleting chemotherapy, JCAR014 infusion or durvalumab infusion
* History of solid organ transplantation

EXCLUSION CRITERIA FOR LYMPHODEPLETION CHEMOTHERAPY, JCAR014 AND DURVALUMAB:

* For lymphodepletion chemotherapy, JCAR014 and durvalumab: Subjects with known active CNS involvement by malignancy; subjects with prior CNS disease that has been effectively treated will be eligible if treatment was completed at least 3 months prior to enrollment and there is no evidence of disease or stable abnormalities on repeat imaging
* Uncontrolled infection
* Receipt of live, attenuated vaccine within 28 days prior to the first dose of durvalumab (Note: enrolled patients should not receive live vaccine during the study and for 180 days after the last dose of durvalumab)
* Planned use of corticosteroids (> 10 mg/day prednisone or equivalent) or other systemic immunosuppression is not permitted within 72 hours prior to JCAR014 infusion; topical and/or inhaled steroids are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Gauthier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Hirayama AV, Kimble EL, Wright JH, Fiorenza S, Gauthier J, Voutsinas JM, Wu Q, Yeung CCS, Gazeau N, Pender BS, Kirchmeier DR, Torkelson A, Chutnik AN, Cassaday RD, Chapuis AG, Green DJ, Kiem HP, Milano F, Shadman M, Till BG, Riddell SR, Maloney DG, Turtle CJ. Timing of anti-PD-L1 antibody initiation affects efficacy/toxicity of CD19 CAR T-cell therapy for large B-cell lymphoma. Blood Adv. 2024 Jan 23;8(2):453-467. doi: 10.1182/bloodadvances.2023011287. PMID 37903325
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was enrolled on the trial but did not move on to treatment. They were not assigned to an arm or to a treatment dose level.
Groups:
- Group I (JCAR014, Durvalumab) Late- Dose Level 1: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - late: start durvalumab no earlier than 21 days after JCAR014
  Group 1 Dose Level 1 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
Period: Overall Study
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Started | 5 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Completed | 1 | 1 | 3 | 0 | 1 | 2 | 3 | 1
Not Completed | 4 | 2 | 0 | 1 | 0 | 1 | 3 | 6
Not completed — Death | 3 | 2 | 0 | 1 | 0 | 0 | 3 | 4
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pt moved to new therapy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5 | Total
Number analyzed (Participants) | 5 | 3 | 3 | 1 | 1 | 3 | 6 | 7 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2 | 1 | 0 | 3 | 5 | 4 | 17
  >=65 years | 3 | 3 | 1 | 0 | 1 | 0 | 1 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 0 | 1 | 3 | 3 | 10
  Male | 3 | 3 | 2 | 1 | 1 | 2 | 3 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 3 | 1 | 1 | 3 | 6 | 7 | 28
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 5 | 2 | 3 | 1 | 1 | 3 | 4 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Who Experienced Adverse Events
Description: Toxicity graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03.
Time Frame: 28 days post last infusion of Durvalumab, up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Group I (JCAR014, Durvalumab) Early - Dose Level 2: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - early: start durvalumab no earlier than 7 days after JCAR014.
  Group 1 Dose Level 1 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
- Group I (JCAR014, Durvalumab) Late- Dose Level 1: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - late: start durvalumab no earlier than 21 days after JCAR014
  Group 1 Dose Level 2 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
  .
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
- Group I (JCAR014, Durvalumab) Late - Dose Level 2: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - late: start durvalumab no earlier than 21 days after JCAR014
  Group 1 Dose Level 2 is 750 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
- Group II (Durvalumab, JCAR014) - Dose Level 1: Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 1 is 7.5 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
- Group II (Durvalumab, JCAR014) - Dose Level 2: Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 2 is 22.5 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
- Group II (Durvalumab, JCAR014) - Dose Level 3: Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 3 is 75 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
- Group II (Durvalumab, JCAR014) - Dose Level 4: Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 4 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
- Group II (Durvalumab, JCAR014) - Dose Level 5: Patients receive durvalumab IV over 60 minutes on day -1, JCAR014 IV over 20-30 minutes on day 0, then up to 10 additional doses of durvalumab every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Group 2 Dose Level 5 is 750 mg Durvalumab, up to 2 x 106/kg CAR T cells
  Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ Central Memory T-lymphocytes JCAR014: Given IV
  Cyclophosphamide: Given IV
  Durvalumab: Given IV
  Fludarabine: Given IV
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 5 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Participants | 5 | 3 | 3 | 1 | 1 | 3 | 6 | 7

2. Primary Outcome: Dose Limiting Toxicity (DLT) Rates
Description: Will be summarized based on the dose limiting toxicity evaluable analysis set. The target toxicity rate for the maximum tolerated dose is 30%. Outcome will be reported as a count of patients in each arm that experienced a DLT.
Time Frame: 28 days post first infusion of Durvalumab (for participants in Group 1) or 28 days post infusion of JCAR (for participants in Group 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 5 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Highest Treatment Dose Administered on Study
Description: Reporting outcome as the maximum durvalumab dose that we reached on the study. Patients were monitored for 28 days post infusion for dose limiting toxicities. The DLT rate was used to determine dose escalation. The study was terminated prior to reaching the maximum tolerated dose.
Time Frame: 28 days
Measure: Number; unit: mg
Groups:
- All Treated Patients: Arm contains all treated patients on study
Arm/Group | All Treated Patients
Number analyzed (Participants) | 29
mg | 750

4. Primary Outcome: Maximum JCAR014 Cmax by Flow Cytometry
Description: Absolute CD4+ and CD8+ CAR-T cell counts were determined by multiplying the percentages of CD3+CD4+CD8-EGFRt+ and CD3+CD4-CD8+EGFRt+ events, respectively, in a viable CD45+ lymphocyte forward/side scatter gate by an absolute lymphocyte count performed on the same day. Excluding 1 patient in Group 2 Dose Level 5 who received an out-of-specification JCAR014 product.
Time Frame: Up to 12 months
Measure: Mean (Full Range); unit: CD3+ CAR-T cells/μL
Groups:
- Group I (JCAR014, Durvalumab) - Dose Level 1: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 Dose Level 1 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
- Group I (JCAR014, Durvalumab) - Dose Level 2: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 Dose Level 2 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
Arm/Group | Group I (JCAR014, Durvalumab) - Dose Level 1 | Group I (JCAR014, Durvalumab) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 3 | 8 | 1 | 1 | 3 | 6 | 6
CD3+ CAR-T cells/μL | 201.21 [9.86 to 555.77] | 13.71 [1.88 to 36.51] | 8.27 [8.27 to 8.27] | 3.01 [3.01 to 3.01] | 13.15 [3.51 to 32.10] | 18.13 [5.16 to 51.49] | 7.53 [1.44 to 13.83]

5. Primary Outcome: Area Under the Curve (AUC) of JCAR014 by Flow Cytometry
Description: Absolute CD4+ and CD8+ CAR-T cell counts were determined by multiplying the percentages of CD3+CD4+CD8-EGFRt+ and CD3+CD4-CD8+EGFRt+ events, respectively, in a viable CD45+ lymphocyte forward/side scatter gate by an absolute lymphocyte count performed on the same day. Subjects had samples analyzed at approximately days 0, 3, 7, 10, 14, 21, and 28 after CAR-T cell infusion to generate the AUC from day 0 to 28. The areas under the curve of CAR T-cell counts by flow cytometry and qPCR between time points were calculated by using a trapezoidal rule computational algorithm. Excluding 1 patient in Group 2 Dose Level 5 who received an out-of-specification JCAR014 product.
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: Days x CD3+ CAR-T cells/μL
Arm/Group | Group I (JCAR014, Durvalumab) - Dose Level 1 | Group I (JCAR014, Durvalumab) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 3 | 8 | 1 | 1 | 3 | 6 | 6
Days x CD3+ CAR-T cells/μL | 844.77 [105.13 to 2078.77] | 104.33 [10.01 to 316.62] | 47.96 [47.96 to 47.96] | 32.44 [32.44 to 32.44] | 90.78 [23.13 to 220.87] | 160.94 [54.43 to 330.53] | 71.97 [14.39 to 162.37]

6. Primary Outcome: Maximum JCAR014 Cmax in Blood by Quantitative Polymerase Chain Reaction (qPCR) Analysis
Description: The number of copies of the CAR transgene/μg of DNA in the blood was determined by using quantitative polymerase chain reaction (qPCR) to detect the integrated Flap-EF1⍺ sequence, with a lower limit of detection of 10 transgene copies/μg of DNA. Excluding 1 patient in Group 2 Dose Level 5 who received an out-of-specification JCAR014 product.
Time Frame: Up to 12 months
Measure: Mean (Full Range); unit: CAR transgene copies/μg DNA
Arm/Group | Group I (JCAR014, Durvalumab) - Dose Level 1 | Group I (JCAR014, Durvalumab) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 3 | 8 | 1 | 1 | 3 | 6 | 6
CAR transgene copies/μg DNA | 37647.95 [3699.84 to 97951.33] | 10043.68 [1717.18 to 25286.16] | 3690.24 [3690.24 to 3690.24] | 1949.22 [1949.22 to 1949.22] | 8295.36 [1120.19 to 20755.61] | 27841.31 [1927.33 to 87193.83] | 26297.43 [1515.33 to 122322.41]

7. Primary Outcome: AUC of JCAR014 Cells by qPCR Analysis
Description: The number of copies of the CAR transgene/μg of DNA in the blood was determined by using quantitative polymerase chain reaction (qPCR) to detect the integrated Flap-EF1⍺ sequence, with a lower limit of detection of 10 transgene copies/μg of DNA. Subjects had samples analyzed at approximately days 0, 3, 7, 10, 14, 21, and 28 after CAR-T cell infusion to generate the AUC from day 0 to 28.The areas under the curve of CAR T-cell counts by flow cytometry and qPCR between time points were calculated by using a trapezoidal rule computational algorithm. Excluding 1 patient in Group 2 Dose Level 5 who received an out-of-specification JCAR014 product.
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: CAR transgene copies/μg DNA x days
Arm/Group | Group I (JCAR014, Durvalumab) - Dose Level 1 | Group I (JCAR014, Durvalumab) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 3 | 8 | 1 | 1 | 3 | 6 | 7
CAR transgene copies/μg DNA x days | 296188.95 [40685.13 to 730201.08] | 104088.38 [19729.18 to 433057.46] | 18710.77 [18710.77 to 18710.77] | 16721.68 [16721.68 to 16721.68] | 63778.63 [11246.81 to 155355.19] | 353471.10 [27198.84 to 1266668.39] | 389065.24 [14387.21 to 1811692.73]

8. Primary Outcome: Time to Loss of JCAR014 Detection in Blood by qPCR Analysis
Description: as for outcome 6
Time Frame: Up to 12 months, +/- 30 days
Population: Participants analyzed are the participants with documented loss of detection of JCAR014 in blood by qPCR during follow-up.
Measure: Mean (Full Range); unit: days
Arm/Group | Group I (JCAR014, Durvalumab) - Dose Level 1 | Group I (JCAR014, Durvalumab) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 2 | 3 | 1 | 0 | 3 | 2 | 2
days | 113 [91 to 134] | 191 [49 to 392] | 28 [28 to 28] |  | 199 [168 to 227] | 183 [149 to 217] | 64 [39 to 88]

9. Secondary Outcome: Rate of Complete Response (CR) by Investigator Assessment Using Lugano Criteria
Description: This outcome is a count of participants who experienced a best response of complete response (CR) by investigator assessment using Lugano criteria. 1 patient in Group 1 Early Dose Level 2 could not be analyzed for the outcome because they expired before their first response assessment.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 4 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Participants | 1 | 1 | 2 | 0 | 1 | 2 | 2 | 1

10. Secondary Outcome: Rate of Partial Response (PR) by Investigator Assessment Using Lugano Criteria
Description: This outcome is a count of participants who experienced a best response of partial response (PR) by investigator assessment using Lugano criteria. 1 patient in Group 1 Early Dose Level 2 could not be analyzed for the outcome because they expired before their first response assessment.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 4 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Participants | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1

11. Secondary Outcome: Objective Response Rate by Investigator Assessment Using Lugano Criteria
Description: ORR, defined as a count of participant with a best response of either complete response or partial response. 1 patient in Group 1 Early Dose Level 2 could not be analyzed for the outcome because they expired before their first response assessment.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 4 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Participants | 1 | 1 | 2 | 0 | 1 | 2 | 2 | 2

12. Secondary Outcome: Duration of Response
Description: Duration of response will be an average amount of days from first response assessment until progression or death for treated patients. Total number analyzed will be the patients that progressed or died, excluding those that did not progress or die. 1 patient in Group 1 Early Dose Level 2 could not be analyzed for the outcome because they expired before their first response assessment.
Time Frame: From first response to progressive disease or death, assessed up to 1 year
Population: Total number analyzed will be the patients that progressed or died, excluding those that did not progress or die. 1 patient in Group 1 Early Dose Level 2 could not be analyzed for the outcome because they expired before their first response assessment.
Measure: Mean (Full Range); unit: days
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 2 | 2 | 2 | 0 | 1 | 1 | 4 | 7
days | 72.5 [0 to 145] | 47.5 [0 to 95] | 42 [0 to 84] |  | 35 [35 to 35] | 31 [31 to 31] | 97.75 [0 to 357] | 18.14 [0 to 99]

13. Secondary Outcome: Progression Free Survival
Description: Outcome will be reported as a count of those who did not progress and did not die while on study.
Time Frame: From date of first study treatment to progressive disease or death, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 5 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Participants | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 0

14. Secondary Outcome: Overall Survival
Description: Outcome will be reported as a count of participants who survived while on study. Survival was assessed up to 1 year.
Time Frame: From date of first study treatment to death, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late- Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
Number analyzed (Participants) | 5 | 3 | 3 | 1 | 1 | 3 | 6 | 7
Participants | 2 | 1 | 3 | 0 | 1 | 3 | 3 | 3

15. Other Pre Specified Outcome: B-cell Depletion in Circulation, Profile of Soluble Circulating Proteins Such as Cytokines and Chemokines, and Changes in the Level of Detectable Soluble PD-L1
Time Frame: Up to 12 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in the Phenotype of Tumor Cells (e.g., Expression of PD-L1) and of the Tumor Microenvironment (e.g., Infiltration by Chimeric Antigen Receptor [CAR] T Cells)
Description: Flow cytometry may be used in the blood, bone marrow, and cerebrospinal fluid (CSF) (if applicable).
Time Frame: Baseline up to 12 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Phenotype and/or Genetic Profile of Endogenous Immune Cells and CAR T Cells
Description: Flow cytometry may be used in the blood, bone marrow, and CSF (if applicable).
Time Frame: Up to 12 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Cmax of Durvalumab in Serum
Time Frame: Up to 12 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: AUC of Durvalumab in Serum
Time Frame: Up to 12 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Clearance of Durvalumab in Serum
Time Frame: Up to 12 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Terminal Half-life of Durvalumab in Serum
Time Frame: Up to 12 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Antibodies and Cellular Immune Responses to JCAR014
Description: Cellular immune responses to JCAR014 will be considered in patients who have two consecutive negative assays for JCAR014 or who have recovered endogenous B cells. Cellular responses to JCAR014 will be evaluated by assessing reactivity of patient peripheral T cells to JCAR014. Peripheral blood will be collected for these studies.
Time Frame: Up to 12 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Anti-drug Antibodies Directed Against Durvalumab
Description: Will be assessed using a validated immunoassay in serum samples.
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 days post last infusion of Durvalumab, up to 1 year
Description: An adverse event (AE) is the development of any untoward medical occurrence or the clinical deterioration of a pre-existing medical condition in a patient or clinical study patient administered a medicinal product (e.g., JCAR014 and/or durvalumab). Reporting of AEs will be based on the Medical Dictionary for Regulatory Activities (MedDRA) and CTCAE version 4.03.
Groups:
- Group I (JCAR014, Durvalumab) Early - Dose Level 2: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - early: start durvalumab no earlier than 7 days after JCAR014.
  Group 1 Dose Level 1 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
- Group I (JCAR014, Durvalumab) Late - Dose Level 1: Patients receive JCAR014 IV over 20-30 minutes on day 0 and durvalumab IV over 60 minutes on day 21 (may occur as early as day 7) and then every 4 weeks for up to 10 doses in the absence of disease progression or unacceptable toxicity.
  Group 1 - late: start durvalumab no earlier than 21 days after JCAR014
  Group 1 Dose Level 2 is 225 mg Durvalumab, up to 2 x 106/kg CAR T cells
Arm/Group | Group I (JCAR014, Durvalumab) Early - Dose Level 2 | Group I (JCAR014, Durvalumab) Late - Dose Level 1 | Group I (JCAR014, Durvalumab) Late - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 1 | Group II (Durvalumab, JCAR014) - Dose Level 2 | Group II (Durvalumab, JCAR014) - Dose Level 3 | Group II (Durvalumab, JCAR014) - Dose Level 4 | Group II (Durvalumab, JCAR014) - Dose Level 5
All-Cause Mortality (participants affected / at risk) | 3/5 | 2/3 | 0/3 | 1/1 | 0/1 | 0/3 | 3/6 | 4/7
Serious Adverse Events (participants affected / at risk) | 4/5 | 3/3 | 2/3 | 1/1 | 0/1 | 2/3 | 4/6 | 4/7
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3 | 1/1 | 1/1 | 3/3 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (JCAR014, Durvalumab) Early - Dose Level 2 (N=5) | Group I (JCAR014, Durvalumab) Late - Dose Level 1 (N=3) | Group I (JCAR014, Durvalumab) Late - Dose Level 2 (N=3) | Group II (Durvalumab, JCAR014) - Dose Level 1 (N=1) | Group II (Durvalumab, JCAR014) - Dose Level 2 (N=1) | Group II (Durvalumab, JCAR014) - Dose Level 3 (N=3) | Group II (Durvalumab, JCAR014) - Dose Level 4 (N=6) | Group II (Durvalumab, JCAR014) - Dose Level 5 (N=7)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DUODENAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FEVER (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
BACTEREMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: CENTRAL LINE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: COAG NEGATIVE STAPHYLOCOCCUS BACTEREMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER,SPECIFY: PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (JCAR014, Durvalumab) Early - Dose Level 2 (N=5) | Group I (JCAR014, Durvalumab) Late - Dose Level 1 (N=3) | Group I (JCAR014, Durvalumab) Late - Dose Level 2 (N=3) | Group II (Durvalumab, JCAR014) - Dose Level 1 (N=1) | Group II (Durvalumab, JCAR014) - Dose Level 2 (N=1) | Group II (Durvalumab, JCAR014) - Dose Level 3 (N=3) | Group II (Durvalumab, JCAR014) - Dose Level 4 (N=6) | Group II (Durvalumab, JCAR014) - Dose Level 5 (N=7)
ANEMIA (Blood and lymphatic system disorders) | 2 (2) | 2 (10) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 4 (10) | 4 (12)
INVESTIGATIONS - OTHER, SPECIFY: INCREASED NUCLEATED RED BLOOD CELLS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (6) | 3 (13) | 0 (0) | 2 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 3 (4) | 2 (27) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 6 (13) | 4 (8)
SINUS TACHYCARDIA (INTERMITTENT) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA, INTERMITTENT (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY: CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLURRED VISION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY: PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLOATERS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (19) | 2 (3) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 1 (1)
ABDOMINAL PAIN (AND DISCOMFORT) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN, INTERMITTENT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOATING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 3 (9) | 3 (3) | 1 (1) | 1 (3) | 2 (2) | 5 (6) | 4 (9)
CONSTIPATION, INTERMITTENT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (3) | 4 (5) | 2 (2)
DIARRHEA, INTERMITTENT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
DUODENAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
DYSPHAGIA (INCREASED) (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY: GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERMITTENT ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTERMITTENT DIARRHEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (3) | 3 (13) | 2 (4) | 0 (0) | 1 (1) | 3 (12) | 5 (8) | 5 (9)
NAUSEA (INTERMITTENT) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA, INTERMITTENT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 1 (2) | 4 (7)
VOMITTING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
WORSENING OF CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRUISING (INJECTION SITE) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRUISING (PICC SITE) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
EDEMA (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EDEMA LIMBS (General disorders) | 0 (0) | 2 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (6)
EDEMA TRUNK (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
FATIGUE (General disorders) | 4 (17) | 3 (11) | 3 (9) | 0 (0) | 1 (1) | 3 (11) | 6 (17) | 6 (20)
FATIGUE (INTERMITTENT) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE, INTERMITTENT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FEVER (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLU-LIKE SYMPTOMS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY: RIGORS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY: COLD SENSATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY: NODULE ON L SOLE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY: TROUBLE GETTING WARM (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENERAL DISORDERS AND SITE ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY: TIGHTNESS IN CHEST (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
GENERALIZED BODY PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: HICKMAN LINE RASH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: PORT RASH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: PORT SITE IRRITATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: REDNESS AT PICC SITE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MILD ERYTHEMA AND PRURITUS UNDER HICKMAN DRESSING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — INJURY, POISONING, AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY
INTERMITTENT FEVERS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY: EARLY SATIETY (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PORT SITE IRRITATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PORT SITE PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIGORS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: ERYTHEMA AT HICKMAN SITE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: HICKMAN LINE RASH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: HICKMAN LINE RASH, INTERMITTENT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: LINE BANDAGE SITE BLISTER (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: PICC RASH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: PIV RASH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY: CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY: GALLSTONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY: HYPOGAMMAGLOBULINEMIA (Immune system disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
IMMUNE SYSTEMS DISORDERS- OTHER, SPECIFY: HYPOGAMMAGLOBULINEMIA (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: BACTEREMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: CENTRAL LINE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: ORAL THRUSH (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: PARAINFLUENZA 2 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: PARAINFLUENZA 4 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: RESPIRATORY SYNCYTIAL VIRUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER,SPECIFY: BACTEREMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: HICKMAN SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
MUCOSAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARANGEAL CANDIDIASIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAPULOPUSTULAR RASH (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHINOVIRUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
VASCULAR DISORDERS - OTHER, SPECIFY: SEPTIC PULMONARY EMBOLI (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 3 (3)
BRUISING, INTERMITTENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS RADIATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: FLEA BITES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: BIOPSY SITE PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: PAIN AT BIOPSY SITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: PAIN FROM BONE MARROW ASPIRATE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: TORN MENISCUS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INJURY, POISONING, AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY: CUT ON LEFT FINGER (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY: FINGER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY: SYSTOLIC MURMUR (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CARDIAC TROPONIN I INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED NEUTROPHIL COUNT (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBRINOGEN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FIBROGEN COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: ASTROVIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (3) | 3 (8) | 3 (12) | 1 (1) | 1 (5) | 3 (12) | 6 (14) | 5 (21)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 1 (8) | 1 (1) | 0 (0) | 1 (6) | 0 (0) | 1 (1) | 4 (17)
WEIGHT GAIN (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
WEIGHT LOSS (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 3 (5) | 3 (10) | 1 (2) | 0 (0) | 1 (1) | 1 (4) | 5 (12) | 4 (7)
ANOREXIA (INTERMITTENT) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANOREXIA, INTERMITTENT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (7)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (3) | 0 (0) | 1 (1) | 3 (10) | 3 (4)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 2 (3)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
INVESTIGATIONS - OTHER, SPECIFY: HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INVESTIGATIONS - OTHER, SPECIFY: IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
INVESTIGATIONS -OTHER, SPECIFY: IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY: HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY: TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY: GOUT PAIN (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY: GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
ARTHRALGIA, INTERMITTENT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 1 (1) | 3 (7)
BILATERAL KNEE JOINT PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY: HIP BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 2 (2)
GENERALIZED MUSCLED WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEFT LEG BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE - OTHER, SPECIFY: LEFT WRIST TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY: RIGHT HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: BACK STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: EXERCISE INDUCED MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: JAW PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: JOINT PAIN DUE TO GARDENING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: MUSCLE SORENESS AFTER ACTIVITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: MYALGIA AFTER EXERCISE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: RIGHT FOOT PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - OTHER, SPECIFY: SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN, INTERMITTENT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RIB PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WORSENING OF LLQ BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS SKIN DISORDERS - OTHER, SPECIFY: BASAL CELL LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 3 (8)
COGNITIVE DISTURBANCE (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (3) | 2 (9) | 1 (1) | 0 (0) | 1 (1) | 3 (6) | 2 (3) | 3 (6)
DIZZINESS (INTERMITTENT) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS, INTERMITTENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
EYE DISORDERS - OTHER, SPECIFY: HORNER'S SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY: HYPEROSMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 4 (9)
HEADACHE, INTERMITTENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERSOMNIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERMITTENT DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERMITTENT PARESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LETHARGY, INTERMITTENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY: MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY: ULNAR NERVE FINGER NUMBESS WITH SHOULDER ABDUCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARATHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL NEUROPATHY (HANDS) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL NEUROPATHY, INTERMITTENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (3) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY, INTERMITTENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
TREMORS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 3 (4)
ANXIETY, INTERMITTENT (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
CONFUSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
INSOMNIA (Psychiatric disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 4 (7)
INSOMNIA (INTERMITTENT) (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA, INTERMITTENT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INTERMITTENT ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERMITTENT INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY: FLAT AFFECT (Psychiatric disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEMATURIA, INTERMITTENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY: DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY: HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY: NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL AND URINARY DISORDERS - OTHER,SPECIFY: NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
RENAL CALCULI (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1)
URINARY HESITANCY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENITAL EDEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY: BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY: NIPPLE PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER,SPECIFY: VAGINAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALLERGIC RHINITIS, INTERMITTENT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ALLERGIC RHITINITIS, INTERMITTENT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 3 (3) | 3 (4) | 2 (4)
DSYPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (6) | 3 (4) | 0 (0) | 1 (4) | 1 (1) | 4 (7) | 3 (7)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
INTERMITTENT COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
NASAL CONGESTION, INTERMITTENT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (3)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY: TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY: BRADYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY: HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
BULLOUS DERMITITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIAPHORESIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
DRY SKIN INTERMITTENT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN, INTERMITTENT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOREHEAD PRURITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RASH (BILATERAL FLANKS AND BACK) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
RASH MACULOPAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (4)
SKIN AND SUBCUTANEOUS CONDITIONS - OTHER, SPECIFY: LOCALIZED ERYTHEMA OF THE NECK (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - LIVEDO RETICULARIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: DIAPHORESIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: HEAT RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: INGROWN TOENAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: NIGHT SWEATS, INTERMITTENT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY: VENOUS STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN NODULE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY: NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HOT FLASHES (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (6) | 0 (0) | 2 (4) | 1 (1) | 1 (5) | 2 (11) | 4 (13) | 5 (16)
HYPERTENSION, INTERMITTENT (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 3 (5) | 3 (27) | 2 (2) | 0 (0) | 1 (7) | 3 (8) | 5 (12) | 4 (6)
HYPOTENSION, INTERMITTENT (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RIGHT LEG LYMPHEDEMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT02706405/Prot_SAP_000.pdf